CLINICAL TRIAL: NCT03782207
Title: A Non-Interventional, Multicenter, Multiple Cohort Study Investigating the Outcomes and Safety of Atezolizumab Under Real-World Conditions in Patients Treated in Routine Clinical Practice
Brief Title: A Study Investigating the Outcomes and Safety of Atezolizumab Under Real-World Conditions in Patients Treated in Routine Clinical Practice
Acronym: IMreal
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO40653
Record Dates: First submitted 2018-11-28; First posted 2018-12-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma; Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Cohort 1 (UC LOT2+later lines[LOT2+] & platinum eligible LOT1): Participants diagnosed with locally advanced or metastatic Urothelial Cancer previously treated with platinum-containing chemotherapy.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab
- Cohort 2 (NSCLC LOT2 plus later lines [LOT2+]): Participants diagnosed with Locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) after prior chemotherapy. Participants with epidermal growth factor receptor (EGFR) activating mutations or anaplastic lymphoma kinase (ALK)-positive tumor mutations should also have received targeted therapy.
  Enrollment closed.
  Interventions: Drug: Atezolizumab
- Cohort 3 (NSCLC LOT1 plus EGFR+/ALK+ LOT2+): EMA: Participants diagnosed with locally advanced/metastatic non-squamous NSCLC not previously treated. Participants with EGFR-activating mutations or ALK-positive tumor mutations should have received at least one line of targeted therapy.
  FDA: for the treatment of adult participants with metastatic NSCLC who have disease progression during or following platinum-containing chemotherapy. Participants with EGFR or ALK genomic tumor aberrations should have disease progression on FDA-approved therapy for NSCLC harboring these aberrations prior to receiving TECENTRIQ.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab
- Cohort 4 (ES-SCLC LOT1): Participants diagnosed with extensive stage (ES) small cell lung cancer (SCLC) not previously treated.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab
- Cohort 5 (NSCLC LOT1): Participants diagnosed with metastatic Non-Small Cell Lung cancer with high PD-L1 expression, previously untreated.
  Interventions: Drug: Atezolizumab
- Cohort 6 (HCC LOT1): Participants diagnosed with unresectable locally advanced or metastatic hepatocellular carcinoma previously untreated with systemic therapy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at the discretion of the treating physician per local guidelines and independently of participation in this study.
  Other Names: Tecentriq

SUMMARY:
This is a non-interventional, multi-country, multi-centre, multiple cohort prospective study, with retrospective collection of prior medical/treatment history data from medical records, designed to assess the real-world outcomes and safety of atezolizumab for indications in the existing label in the real world setting of routine clinical practice.

DETAILED DESCRIPTION:
The study will be split into separate cohorts based on the approved indications for atezolizumab treatment, excluding cisplatin ineligible participants receiving atezolizumab as first line of therapy (LOT1) for locally advanced/metastatic urothelial cancer (locally advanced/metastatic UC). The study may be amended for inclusion of new cohorts as these are approved in the participating countries. Participants will be included into each cohort based on their indication for receiving atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have one of the following confirmed diagnoses for which atezolizumab is locally approved in the SmPC: (1) As monotherapy for the treatment of adult patients with locally advanced/metastatic UC after prior platinum-containing chemotherapy (Cohort 1 LOT2+mUC) or (2) As monotherapy for the treatment of adult patients with locally advanced/metastatic NSCLC after prior chemotherapy. Patients with EGFR activating mutations or ALK-positive tumour mutations should also have received targeted therapy before receiving atezolizumab (Cohort 2 LOT2+NSCLC) or (3) In combination with bevacizumab, paclitaxel and carboplatin for the first line treatment of adult patients with metastatic non-squamous NSCLC. Patients with EGFR activating mutations or ALK- positive tumour mutations should also have received targeted therapy (Cohort 3 LOT1 NSCLC) or (4) In combination with carboplatin and etoposide, is indicated for the first-line treatment of adult patients with extensive-stage small cell lung cancer (ES-SCLC) (Cohort 4 LOT1 ES-SCLC) or (5) As a monotherapy, for the treatment of metastatic NSCLC with high PD-L1 expression, previously untreated (Cohort 5 LOT1 NSCLC) or (6) In combination with bevacizumab for unresectable locally advanced or metastatic hepatocellular carcinoma previously untreated with systemic therapy (Cohort 6 LOT1 HCC) .
* Patient is administered atezolizumab therapy for the first time.
* Decision to administer atezolizumab must be made and documented prior to inclusion into the study and must follow local clinical practice.

Exclusion Criteria:

* Patients not receiving treatment for a disease with atezolizumab according to standard of care and in line with the current summary of product characteristics (SPC) or local labelling. Cisplatin ineligible patients receiving atezolizumab LOT1 for the treatment of locally advanced/metastatic UC patients will be excluded
* Concomitant anti-cancer therapy at the time of starting atezolizumab on the index date not part of locally approved combination therapy with atezolizumab.
* Treatment with atezolizumab as part of a clinical trial or for compassionate use as part of a pre-approval or compassionate use program.
* Patients not receiving atezolizumab, but a biosimilar or non-original biologic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with locally advanced /mUC previously treated with platinum-containing chemotherapy, participants diagnosed with locally advanced/metastatic non-small cell lung cancer (NSCLC) after prior chemotherapy, participants diagnosed with extensive-stage small cell lung cancer (ES-SCLC), participants diagnosed with metastatic NSCLC previously untreated,and participants diagnosed with locally unresectable locally advanced or metastatic hepatocellular carcinoma previously untreated with systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2756 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Index date up to approximately 6 years
  Time from index date until date of death from any cause. Index date is the date of administration of the first ever dose of atezolizumab for each patient.
OS at 2 Years | After index date up to 2 years
  Percentage of participants alive 2 years after initiation of atezolizumab treatment.

SECONDARY OUTCOMES:
Time to Loss of Clinical Benefit (TTLCB) | Index date up to approximately 6 years
  Time from the index date to loss of clinical benefit as assessed by the treating physician.
Progression Free Survival (PFS) | Index date up to approximately 6 years
  Time from index date to death or disease progression (PD).
Objective Response Rate (ORR) | After index date up to approximately 6 years
  Percentage of participants who have a best overall response (BOR) of Complete Response (CR) or Partial Response (PR). BOR for each participant is the best response achieved after the index date prior to initiation of any subsequent treatment.
Time to Response | Index date up to approximately 6 years
  Time from index date to first objective tumor response, CR or PR.
Duration of Response (DoR) | Index date up to approximately 6 years
  Time from first documentation of CR or PR (whichever occurs first) after index until death or PD.
Disease Control Rate (DCR) | From 12 weeks after index date up to approximately 6 years
  Percentage of participants who have achieved CR, PR and stable disease at least 12 weeks after the index date.
Duration of DCR | After index date up to approximately 6 years
  Time from first documentation of CR, PR or stable disease (whichever occurs first) after index until death or PD.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire Score | Index date or after ICF signature, & approx. at 6, 12, and 24 weeks of treatment; then at approx. 3 months, 6 months, 12 months, & every 12 months thereafter until end of study (study planned duration up to approximately 6 years)
  EQ-5D-5L during and after atezolizumab treatment will be used to assess HRQoL. Scale is from 1-5 (no problems, slight problems, moderate problems, severe problems and extreme problems).
Number of Paricipants with Disease Stage TNM and IUCC | At index date (Index date is the date of administration of the first ever dose of atezolizumab for each patient.)
Number of Participants at Each Level of Karnofsky or ECOG Performance Status | At index date (Index date is the date of administration of the first ever dose of atezolizumab for each patient.
Total Number of Infusions of Atezolizuamb | Treatment period until discontinuation (up to approximately 6 years)
Duration of Treatment With Atezolizumab | Index date until date of treatment discontinuation (up to approximately 6 years)
Time to initiation of the first subsequent cancer-related therapy | Up to approximately 6 years
Percentage of Participants with Adverse Events | Up to approximately 6 years
Number of Lines of Prior and Subsequent Cancer-Related Therapies | Up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (258):
- Argentina (7):
  - Hospital Universitario Austral, Buenos Aires
  - Lucen S.A., Buenos Aires
  - Consultorio Privado Korbenfeld, CABA
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Sanatorio de la Mujer, Rosario
  - Fundacion Koriza, Santa Rosa
- Austria (4):
  - Klinikum Klagenfurt, Klagenfurt
  - Landesklinikum Krems, Krems
  - Salzkammergut-Klinikum Voecklabruck, Vöcklabruck
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (6):
  - AZ KLINA, Brasschaat
  - AZ St Maarten Campus Leopoldstr, Mechelen
  - CHU UCL Mont-Godinne, Mont-godinne
  - AZ Oostende, Ostend
  - AZ Delta (Campus Rumbeke), Roeselare
  - Sint Trudo Ziekenhuis, Sint-Truiden
- Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo, Brazil
- Bulgaria (13):
  - Complex Oncology Center Burgas, Burgas
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
  - Umhat Dr Georgi Stranski, Pleven
  - University Hospital Palmed, Plovdiv
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - Complex Oncology Center - Plovdiv First Internal Chemotherapy Department, Plovdiv
  - DDODIU-Plovdiv, EOOD, Plovdiv
  - Complex Oncological Center-Ruse EOOD, Rousse
  - Tokuda Hospital, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MBAL Serdika EOOD, Sofia
  - MHAT SofiaMed, Sofia
  - Specialized Hospital for Active Cancer Treatment, Dr. Mark Antonov Markov - Varna Ltd, Varna
- Centro de Estudios Clínicos SAGA, Santiago, Chile
- Colombia (4):
  - Angiografia del Occidente, Cali
  - Fundacion Clinica Valle del Lili, Cali
  - Hospital Pablo Tobon Uribe, Medellín
  - Clinica ASTORGA, Medellín
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - Klinicki Bolnicki Centar Split, Split
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Egypt (6):
  - SUN Oncology center- Alexandria, Alexandria
  - Yasser Abdel Kader Private Clinic, Cairo
  - Air Force Specialized Hospital, Cairo
  - Barsoum Oncology Center, Cairo
  - Cairo Oncology Center, Cairo
  - International Medical Center, Cairo
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu Uni Hospital, Tartu
- France (52):
  - Clinique Du Docteur Calabet, Agen
  - Ch Du Pays D Aix, Aix-en-Provence
  - Clinique de l'Europe, Amiens
  - Centre Hospitalier Uni Ire, Angers
  - Hopital Prive D Antony, Antony
  - CHG Henri Dufaut médecine interne-onco-hematologie, Avignon
  - CH de Beauvais, Beauvais
  - Hopital Jean Minjoz, Besançon
  - Ch De Beziers, Béziers
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Cote De Nacre, Caen
  - Ch De Chambery, Chambéry
  - Oncologie 37, Chambray-lès-Tours
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Ch De Compiegne, Compiègne
  - Ch Laennec, Creil
  - Centre Georges Francois Leclerc, Dijon
  - Hopital Simone Veil Eaubonne, Eaubonne
  - Chi Alpes Du Sud Site De Gap, Gap
  - Hopital Nord Ouest, Gleizé
  - Ch Saint Louis, La Rochelle
  - Hopital La Source, La Source
  - Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Du Mans, Le Mans
  - Hôpital Privé La Louviere, Lille
  - Hopital Dupuytren, Limoges
  - Ch Bretagne Sud Site Scorff, Lorient
  - Hopital Privé Jean Mermoz, Lyon
  - Hopital Europeen, Marseille
  - Clinique Clementville, Montpellier
  - Centre Regional de Lutte contre le Cancer Val d Aurelle - Paul Lamarque, Montpellier
  - Hopital Emile Muller, Mulhouse
  - Hopital Caremeau, Nîmes
  - Polyclinique Kenval, Nîmes
  - Institut Curie, Paris
  - Hopital Cochin, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier, Pau
  - Centre Catalan D' Oncologie, Perpignan
  - Ch Annecy - Genevois, Pringy
  - Hopital De La Maison Blanche, Reims
  - Clinique Mutualiste L Estuaire, Saint-Nazaire
  - Hopital Nord, Saint-Priest-en-Jarez
  - Ch De Saint Quentin, Saint-Quentin
  - Hopital Robert Pax, Sarreguemines
  - Hopital Sainte Musse, Toulon
  - Hopital Larrey, Toulouse
  - Centre Hospitalier de Valence, Valence
  - Service de pneumologie Clinique médico-chirurgicale Tessier, Valenciennes
  - Ch Bretagne Atlantique, Vannes
  - Hopital Robert Schuman, Vantoux
- Hungary (5):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Semmelweis Egyetem, AOK, Pulmonologiai Klinika, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - University of Pecs, Pécs
  - Református Pulmonológiai Centrum, Törökbálint
- India (7):
  - HCG Cancer Center, Ahmedabad, Gujarat
  - Sunshine Global Hospital (A unit of Baroda Medicare Pvt Ltd), Surat, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - Aster Medcity, Kochi, Kerala
  - MVR Cancer Centre and Research Institute, Kozhikode, Kerala
  - MOC Cancer Care & Research Centre, Mumbai, Maharashtra
  - AIG Hospitals, Gachibowli, Telangana
- Italy (23):
  - Ospedale San Salvatore, UOC Oncologia, L’Aquila, Abruzzo
  - Grande Ospedale Metropolitano, Reggio Calabria, Calabria
  - Az. Osp. Monaldi, Napoli, Campania
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Ospedale S.S. Trinità Nuovo, Sora, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST), Genoa, Liguria
  - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria, Alessandria, Piedmont
  - Ospedale Oncologico A.Businco, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria Di Sassari, Sassari, Sardinia
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima, Catania, Sicily
  - Az. Osp. Uni. Ria Policlinico G. Martino, Messina, Sicily
  - Ospedale Di Macerata, Macerata, The Marches
  - Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Ospedale Nuovo Della Versilia, Lido di Camaiore, Tuscany
  - A.O.U. Integrata Verona - Policlinico G.B. Rossi, Verona, Veneto
  - Azienda ULSS 8 Berica, Vicenza, Veneto
- Kuwait (2):
  - Kuwait Cancer control center, Kuwait City
  - Kuwait Cancer control center, Shuwakh Industrial
- Lebanon (2):
  - Saint George Hospital, Beirut
  - Middle East Institute of Health Hospital, Bsalim, Mount Lebanon-Metn
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Public Institution, Kaunas
  - National Cancer Institute, Vilnius
- Mexico (3):
  - Medica sur Hospital, Mexico City, Mexico CITY (federal District)
  - Clinica Opcion Oncologia S.A. de C.V., Monterrey, Nuevo León
  - Oncare, San Pedro Garza García, Nuevo León
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, locatie Oost, Amsterdam
  - Catharina ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Zaans Medisch Centrum, Zaandam
- Oman (2):
  - Royal Hospital, Muscat
  - Sultan Qaboos Comprehensive Cancer Care & Research Center, Muscat
- Pakistan (2):
  - Shaukat Khanum Memorial Cancer Hospital, Lahore, Punjab Province
  - Aga Khan University, Karachi, Sindh
- Poland (14):
  - WZZOZ Centrum Leczenia Chorob Pluc i Rehabilitacji, ?ód?
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika w ?odzi, ?ód?
  - Beskidzkie Centrum Onkologii - Szpital Miejski im. Jana Pawla II, Bielsko-Bia?a
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Centrum Pulmonologii i Torakochirurgii, Bystra
  - Wojewodzki Szpital Zespolony, Elblag
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego, Grudzi?dz
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu, Późna
  - Instytut Gruzlicy i Chorob P?uc, Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Dolno?L?Skie Centrum Onkologii, Pulmonologii I Hematologii, Wroc?aw
- Portugal (7):
  - Hospital Geral, Coimbra
  - Centro Clinico Champalimaud, Lisbon
  - Hospital Pulido Valente, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - CHVNG/E_Unidade 1, Vila Nova de Gaia
- Romania (2):
  - Institutul Clinic Fundeni Bucuresti, Bucharest
  - Institutul Regional de Gastroenterologie si Hepatologie Prof. Dr. Octavian Fodor, Cluj-Napoca
- Russia (11):
  - Altai Regional Oncological Center, Barnaul, Altayskiy Kray
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky, Krasnoyarsk, Krasnodarskiy Kray
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - Medical Clinic "AB Medical group", Saint Petersburg, Sankt-Peterburg
  - EuroCityClinic, Saint Petersburg, Sankt-Peterburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - SBIH Kaluga Region Clinical Oncology Dispensary, Kaluga
  - Tver Regional Oncology Clinical Dispensary, Tver'
- Tan Tock Seng Hospital, Singapore, Singapore
- Slovenia (3):
  - Institute of Oncology Ljubljana, Ljubljana
  - University Medical Center Ljubljana, Ljubljana
  - Univerzitetni klini?ni center Maribor, Maribor
- Spain (28):
  - Complejo Hospitalario Torrecardenas, Almería, Almeria
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital General de Mataro, Mataró, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complejo Asistencial Universitario De Burgos, Burgos
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital Clinico de Granada, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Quiron de Madrid, Madrid
  - Complejo Hospitalario de Orense, Ourense
  - Hospital General de Segovia, Segovia
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Tawam Hospital, Al Ain City, United Arab Emirates
- United Kingdom (39):
  - Barnet Hospital, Barnet
  - Royal United Hospital, Bath
  - Clatterbridge Cancer Centre, Bebington
  - Queen Elizabeth Hospital, Birmingham
  - Heartlands Hospital, Birmingham
  - East Lancashire Hospitals NHS Trust, Burnley
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Castle Hill Hospital, Cottingham
  - Royal Surrey County Hospital, Guildford
  - Northwick Park Hospital, Harrow
  - Huddersfield Royal Infirmary, Huddersfield
  - Airedale General Hospital, Keighley
  - Royal Marsden Hospital, Kingston upon Thames
  - St James Hospital, Leeds
  - St Bartholomew's Hospital, London
  - Royal Free Hospital, London
  - Guys and St Thomas Hospital, London
  - Queen Elizabeth Hospital, London
  - St George's Hospital, London
  - Royal Marsden Hospital - Fulham, London
  - Hammersmith Hospital, London
  - Charing Cross Hospital, London
  - Maidstone Hospital, Maidstone
  - The Christie, Manchester
  - James Cook Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Weston Park Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Marsden Hospital (Sutton), Sutton
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Pinderfields General Hospital, Wakefield
  - Great Western Hospitals NHS Foundation Trust., Wiltshire
  - New Cross Hospital, Wolverhampton
  - The York Hospital, York

IPD SHARING:
Plan to Share IPD: No